CLINICAL TRIAL: NCT04791748
Title: Validation and Comparison of a Virtual Reality Protocol in Children Without Vestibular Pathology and Children With Chronic Vestibular déficits : Prospective Study ReViCHILD
Brief Title: Virtual Reality in Children With and Without Vestibular Deficits
Acronym: ReViCHILD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP201074; 2020-A02283-36 (Other: ID RCB number)
Record Dates: First submitted 2021-03-02; First posted 2021-03-10 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Vestibular Diseases
Keywords: Chronic vestibular deficit in children; Virtual reality protocol; Multisensory integration; Hand-eye coordination
MeSH Terms: conditions — Vestibular Diseases | interventions — Vestibular Function Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Children and adolescents patients with chronic vestibular deficits (Experimental): Patients aged 7 to 17 years with chronic vestibular deficits
  Interventions: Diagnostic Test: Vestibular tests; Other: Virtual reality
- children and adolescents controls (Active Comparator): Patients aged 7 to 17 years without chronic vestibular deficits
  Interventions: Diagnostic Test: Vestibular tests; Other: Virtual reality
- Adults without chronic vestibular deficits (Active Comparator)
  Interventions: Diagnostic Test: Vestibular tests; Other: Virtual reality
- Adults with chronic vestibular deficits (Active Comparator)
  Interventions: Diagnostic Test: Vestibular tests; Other: Virtual reality

INTERVENTIONS:
Diagnostic Test: Vestibular tests — Screening vestibular test for patients without chronic vestibular deficits Complete vestibular test if not done yet in care of patients with chronic vestibular deficits
Other: Virtual reality — Virtual reality protocol : doing tasks involving hand-eye coordination, in virtual reality, and in different sensory situations

SUMMARY:
Vestibular information is important in establishing a child's static and dynamic postural control. Any vestibular deficit can have major consequences on development, spatial cognition and quality of life.

In order to interact with the world around us, we must simultaneously integrate different sources of sensory informations (vision, hearing, perception of the body...). The brain integrates these different sensory components to form a unified and coherent perception: this is multisensory integration.

Multisensory integration has been studied using virtual reality in adults, in the "spatial orientation" team of the Center for Integrative Neurosciences and Cognition. These experiments were carried out on healthy subjects and in weightless situations (international space station or parabolic flight). However, no protocol has been developed in children or in subjects with vestibular deficit. Virtual reality is interesting for developing such a protocol because it creates multisensory stimulation capable of promoting visual and proprioceptive compensation of the vestibular deficit.

It induces an immersion of the patient in a virtual spatial and temporal environment difficult to carry out with traditional vestibular rehabilitation techniques. Its main advantage is that it is a fun and safe interactive diagnostic and therapeutic tool, which is particularly suitable for children. Being able to modulate certain sensory information using virtual reality, in children without vestibular function deficit and in children with vestibular function deficit, will make it possible to better understand the role of the vestibule in the construction of the self in relation to space and environment. In addition to the scientific aspect, the diagnostic and therapeutic benefits are potentially numerous.

The objective of the study is to determine a reliable, well-tolerated and age-appropriate virtual reality protocol in children without vestibular deficit and in children with chronic vestibular deficit, making it possible to study the hand-eye coordination.

DETAILED DESCRIPTION:
Vestibular information is important in establishing a child's static and dynamic postural control. Any vestibular deficit can have major consequences on development, spatial cognition and quality of life.

In order to interact with the world around us, we must simultaneously integrate different sources of sensory informations (vision, hearing, perception of the body ...). The brain integrates these different sensory components to form a unified and coherent perception: this is multisensory integration.

It is particularly important in children for the acquisition of sitting, standing and then walking. When a congenital vestibular deficit exists, adaptive behaviors using visual and proprioceptive inputs are set up.

Multisensory integration has been studied using virtual reality in adults, in the "spatial orientation" team of the Center for Integrative Neurosciences and Cognition. These experiments were carried out on healthy subjects and in weightless situations (international space station or parabolic flight). However, no protocol has been developed in children or in subjects with vestibular deficit. Virtual reality is interesting for developing such a protocol because it creates multisensory stimulation capable of promoting visual and proprioceptive compensation of the vestibular deficit.

It induces an immersion of the patient in a virtual spatial and temporal environment difficult to carry out with traditional vestibular rehabilitation techniques. Its main advantage is that it is a fun and safe interactive diagnostic and therapeutic tool, which is particularly suitable for children. Being able to modulate certain sensory information using virtual reality, in children without vestibular function deficit and in children with vestibular function deficit, will make it possible to better understand the role of the vestibule in the construction of the self in relation to space and environment. In addition to the scientific aspect, the diagnostic and therapeutic benefits are potentially numerous.

The objective of the study is to determine a reliable, well-tolerated and age-appropriate virtual reality protocol in children without vestibular deficit and in children with chronic vestibular deficit, making it possible to study the hand-eye coordination.

ELIGIBILITY:
Inclusion Criteria:

* Minors aged 7 to 17 years (inclusive)
* Volunteers adult
* Information and consent of holders of parental authority of minors, minors and of adult subjects

Patients :

* Presence of unilateral or bilateral chronic vestibular pathology
* Minor patients followed in consultation at Necker Hospital in the Pediatric ENT department
* Adult patients followed at adult vestibulometry services (Lariboisière and Pitié Salpêtrière Hospitals)

Controls:

* No history of otological surgery and absence of vestibular pathology
* Patients followed in consultation at Necker Hospital, siblings or adult parents

Exclusion Criteria:

* Presence of an ophthalmological pathology (including refractive errors)
* Presence of neurological pathology including epilepsy or any pathology that can alter mobility and interfere with the performance of tasks

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Degree of reproducibility | Day 0
  Doing a task involving hand-eye coordination, in virtual reality, and in different sensory situations. Success rate for each task is measured
Degree of precision | Day 0
  Doing a task involving hand-eye coordination, in virtual reality, and in different sensory situations. Rate of errors during the test

SECONDARY OUTCOMES:
Compare the success rate in eye-hand coordination | Day 0
  Compare eye-hand coordination in :
  * children without vestibular pathology and in children with vestibular déficits.
  * children with vestibular deficits and in adults with vestibular déficits.
  * children without vestibular pathology and in adults without vestibular déficits.
  * adults without vestibular pathology and in adults with vestibular déficits. Success rate for each task will be measured and compared between groups.
Correlate virtual reality results with vestibular test results | Day 0
  Correlation between success rate during virtual reality and vestibular function (normal vestibular function or not in both ears).
Stratify responses to virtual reality by age | Day 0
  Patients without chronic vestibular déficits. Comparison of success rate according to age.
Occurrence of side effects of virtual reality | Day 0
  Possible side effects of virtual reality.
Children's satisfaction concerning the virtual reality protocol | Day 0
  Open satisfaction questionnaire analysis

CONTACTS AND LOCATIONS:
Overall Officials: Françoise Denoyelle, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; François SIMON, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No